CLINICAL TRIAL: NCT02553070
Title: Health Professions Students and Facutly Perceptions of Poisoning Severity
Brief Title: Health Professions Students and Faculty Perceptions of Poisoning Severity
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500799
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Poisoning
MeSH Terms: conditions — Poisoning | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pharmacy Students: Participants will be asked to indicate their perception of poisoning severity by answering a short survey.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Pharmacy students will be asked to participate in a short (5-7 minutes) survey (see below) that contains 21-short cases involving an exposure to a pharmaceutical or non-pharmaceutical agent. All cases involve children less than 19 years of age. Participants will be asked to indicate their year in pharmacy school (1st or 2nd) and their gender (female/male).

SUMMARY:
Inaccurate perceptions of the severity of an exposure may result in unnecessary visits to the Emergency Department or Health Care Facility which can result in crowding of Emergency Departments, unnecessary utilization of valuable health care resources, unnecessary treatments, and or mistakes / errors resulting in harm to the patient.

Inaccurate perceptions about the severity of an exposure can result in delays in proper evaluation and treatment resulting in harm or in some cases death of the patient.

DETAILED DESCRIPTION:
Consumers and health professionals are often surprised about the toxicity (or lack of toxicity) after exposure to a number of pharmaceutical or non-pharmaceutical agents. Past experience with the survey used in this study has indicated that consumers and health professional perform about the same. Most individuals answer less than 50% of questions incorrectly.

Pharmacy students will be asked to participate in a short (5-7 minutes) survey (see below) that contains 21-short cases involving an exposure to a pharmaceutical or non-pharmaceutical agent. All cases involve children less than 19 years of age. Participants will be asked to indicate their year in pharmacy school (1st or 2nd) and their gender (f/m). The survey will be given after a scheduled examination or other classroom activity and will not involve class time. Students will be provided a link to an online version of the survey.

Conclusions will be derived through the analysis of the data. At a later date, all students in the class (whether they participated in the survey or not)students will be provided a link to video that describes the correct answers to each of the cases and an explanation.

ELIGIBILITY:
Inclusion Criteria:

* All pharmacy students who agree to participate

Exclusion Criteria:

* None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pharmacy students in their 1st or 2nd year of pharmacy school.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Survey will be used for perceptions of poisoning severity | Day 1
  Pharmacy students will be asked to participate in a short (5-7 minutes) survey that contains 21-short cases involving an exposure to a pharmaceutical or non-pharmaceutical agent. The survey will consist of two answers, either "Hospital" or "Home". The data will be complied using the percentage of correct answers on the poisoning severity.

CONTACTS AND LOCATIONS:
Overall Officials: Sven A Normann, PharmD, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Pharmacy, Gainesville, Florida, United States